CLINICAL TRIAL: NCT03683472
Title: Developing a Novel Digital Therapeutic for the Treatment of Generalized Anxiety Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MindSciences, Inc. (Industry)
Collaborators: Brown University (Other)
Responsible Party: Principal Investigator, Judson Brewer, Director of Research & Innovation, Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R41MH118130-01 (NIH)
Record Dates: First submitted 2018-06-11; First posted 2018-09-25 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Anxiety Disorders
Keywords: Anxiety, worry, mindfulness, meditation
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (TAU) (No Intervention): Individuals will receive treatment as usual
- TAU and Unwinding Anxiety Phone App (Active Comparator): The Unwinding Anxiety program focuses on teaching individuals 1) to understand how anxious worry is developed and perpetuated through reinforcement learning, 2) how to recognize these worry "habit loops" and 3) how to bring mindful awareness to moments of worry such that they can uncouple feelings of anxiety from reactive worry thinking and "ride out" habitual mind states that perpetuate and reinforce anxiety. Together, these help individuals "unlearn"/extinguish worry at a core mechanistic level.
  Interventions: Behavioral: Unwinding Anxiety Phone App

INTERVENTIONS:
Behavioral: Unwinding Anxiety Phone App — The Unwinding Anxiety program focuses on teaching individuals 1) to understand how anxious worry is developed and perpetuated through reinforcement learning, 2) how to recognize these worry "habit loops" and 3) how to bring mindful awareness to moments of worry such that they can uncouple feelings of anxiety from reactive worry thinking and "ride out" habitual mind states that perpetuate and reinforce anxiety
  Arms: TAU and Unwinding Anxiety Phone App

SUMMARY:
The investigators propose to develop and adapt Unwinding Anxiety phone app specifically for individuals with generalized anxiety disorder.

DETAILED DESCRIPTION:
The study aims are to (1) develop and refine Unwinding Anxiety for individuals with generalized anxiety disorder, (2) determine user engagement and acceptability as well as measure effect sizes of the program vs. treatment as usual, and (3) preliminarily test mechanisms of action. The knowledge gained will set the stage for a number of future studies related to further elucidating the mechanisms of mindfulness, and the clinical efficacy and utility of this type of training delivered via digital therapeutics in general. Specifically, this study will provide necessary variances for powering larger phase 2 studies.

ELIGIBILITY:
Inclusion Criteria:

* Owns a smart phone
* GAD - 7 is equal to or greater than 10

Exclusion Criteria:

* If using psychotropic medication - not on a stable dosage for at least 6 weeks
* Medical disorder of the severity that would interfere with ability to participate
* Not being fluent in English (due to instructions provided in English)
* As needed use (i.e. prn) of benzodiazepines
* Psychotic disorder,
* Previous MT (e.g. MBSR, other Claritas MindSciences training programs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2019-10-17 (Actual)

PRIMARY OUTCOMES:
UA Program engagement | Two months
  Number of modules completed
Change in worry | Baseline, two months
  Penn State Worry Questionnaire (PSWQ)

SECONDARY OUTCOMES:
Change in non-reactivity & awareness | Baseline, two months
  Five Facet Mindfulness Questionnaire - Non-Reactivity subscale (FFMQ)
UA Program Acceptability | Two months
  Net Promoter Score (NPS)

OTHER OUTCOMES:
Change in anxiety | Baseline, two months
  Generalized Anxiety Disorder - 7 items (GAD-7)
Change in self-regulation | Baseline, two months
  Multidimensional Assessment of Interoceptive Awareness (MAIA)

CONTACTS AND LOCATIONS:
Overall Officials: Judson Brewer, Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Taylor VA, Roy A, Brewer JA. Cluster-based psychological phenotyping and differences in anxiety treatment outcomes. Sci Rep. 2023 Feb 21;13(1):3055. doi: 10.1038/s41598-023-28660-7. PMID 36810609
- [Derived] Roy A, Hoge EA, Abrante P, Druker S, Liu T, Brewer JA. Clinical Efficacy and Psychological Mechanisms of an App-Based Digital Therapeutic for Generalized Anxiety Disorder: Randomized Controlled Trial. J Med Internet Res. 2021 Dec 2;23(12):e26987. doi: 10.2196/26987. PMID 34860673

DOCUMENTS (1):
  • Informed Consent Form (2019-05-02): https://cdn.clinicaltrials.gov/large-docs/72/NCT03683472/ICF_000.pdf